CLINICAL TRIAL: NCT06197594
Title: Effects of Proprioceptive Neuromuscular Facilitation Techniques With and Without Rebound Therapy on Trunk Control in Children With Cerebral Palsy
Brief Title: Effects of PNF and Rebound Therapy on Trunk Control in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0739
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy, PNF, Rebound therapy,Trunk Control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive neuromuscular facilitation techniques (Experimental): GROUP A (experimental group)
  PNF based exercises for trunk control duration 45 min 5 session/week for 6 weeks; Resist person concentric contraction while move in sitting .Resist eccentric control as th lie down. Balance using stabilizing reversals or rhythmic stabilization .Resist shoulder pelvis ,head.Trunk exercises dynamic reversals and combination of isotonic to increase trunk strength and coordination .Resist at scapula and lifting combinations for irradiation. Trunk flexion and extension. Reaching forward and to side with return,for this hip flexion, extension ,lateral motion and rotation with the trunk remaining stable Bridging exercises Lower trunk rotation .Weight shifting in long leg sitting
  Interventions: Other: Proprioceptive neuromuscular facilitation techniques
- Rebound Therapy (Active Comparator): Rebound Therapy lying down on trampoline bouncing created.10 times.Hip kneeling bounce and Standing bouncing with physio balls .Jump on trampoline. Learning front drops, seat drops for 5 minutes.
  Resist person concentric contraction while move into sitting .Resist eccentric control as they lie down. Balance using stabilizing reversals to increase trunk stability .Resist shoulder pelvis, head.Trunk exercises: use dynamic reversals and combination of isotonic to increase trunk strength and coordination .Resist at scapula and lifting combination for irradiation. Trunk flexion and extension. Reaching forward and to side with return,for this hip flexion , extension ,lateral motion and rotation with trunk remaining stable Bridging exercises Lower trunk rotation .Weight shifting in long leg sitting
  Interventions: Other: Rebound Therapy

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation techniques — Proprioceptive neuromuscular facilitation techniques
  Arms: Proprioceptive neuromuscular facilitation techniques
Other: Rebound Therapy — Rebound Therapy
  Arms: Rebound Therapy

SUMMARY:
Cerebral palsy is a group of upper motor neuron syndromes with acquired disorders of early brain development .It effects the person's ability to move and maintain balance and posture. It is the most common motor disability of childhood. Proprioceptive neuromuscular facilitation integration pattern stimulates the proprioceptors with in the muscle and tendon to enhance the performance flexibility, balance and helps in trunk mobility. The motor control movement pattern is facilitated by the dynamic and assistive active resistant progressions regaining motor control. Rebound therapy is used to facilitate movement, promote balance, helps in increase or decrease in muscle tone and promotes sensory integration.

This study will evaluate the effects of PNF techniques with and without rebound therapy on trunk control in children with cerebral palsy. It is randomized controlled trial.34 children with cerebral palsy will participate in this study. The participants will be randomized into control group A (n=17) and experimental group (n =17).Only those children will be included who fulfill inclusion criteria. That is both gender, age range 6 to 12 years, having GMFM score of I -II .Those having cognitive and learning difficulties, having age range out of 6 to 12 years. Data will be analyzed through SPSS 29. The control group will practice PNF techniques for trunk control while experimental group will practice rebound therapy along with PNF exercises for trunk control .Both group will receive 45 min session, 5 days a week for 6 weeks. TCMS and TUG scale will be used.

DETAILED DESCRIPTION:
Intervention

GROUP A (experimental group)

After giving baseline therapy experimental group will be given PNF based exercises for trunk control along with rebound therapy .duration will be 45 minutes, 5 session per week for 6 weeks.

PNF exercises will be;

Resist the person's concentric contraction while they move into sitting .Resist the eccentric control as they lie down. Balancing using stabilizing reversals or rhythmic stabilization to increase trunk stability .Resist the shoulder pelvis and head. For Trunk exercises: use dynamic reversals (slow reversals) and combination of isotonic to increase patient trunk strength and coordination .Resist at scapula and lifting combinations to get added irradiation. Trunk flexion and extension. Reaching forward and to the side with return, this requires hip flexion, extension ,lateral motion and rotation with the trunk remaining stable Bridging exercises Lower trunk rotation .Weight shifting in long leg sitting.

REBOUND THERAPY

Rebound therapy session including lying down on trampoline bouncing created by therapist.

It will be 10 repetitions. .Hip kneeling bouncing with physio balls. Standing bouncing with physio balls .Jumping on trampoline. Learning front drops, seat drops, and other function movements will be given for 5 minutes.

GROUP B (control group)

The control group will only be given PNF based trunk exercises. PNF exercises will be; Resist the person's concentric contraction while they move into sitting .Resist the eccentric control as they lie down. Balancing using stabilizing reversals or rhythmic stabilization to increase trunk stability .Resist the shoulder pelvis and head. For Trunk exercises: use dynamic reversals (slow reversals) and combination of isotonic to increase patient trunk strength and coordination .Resist at scapula and lifting combinations to get added irradiation. Trunk flexion and extension. Reaching forward and to the side with return, this requires hip flexion , extension ,lateral motion and rotation with the trunk remaining stable Bridging exercises Lower trunk rotation .Weight shifting in long leg sitting.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Children from 6 years to 12 years of age will be included
* Degree of spasticity ranged from 1 and 1+ according to modified Ashworth scale
* According to gross motor functional classification system children were categorized on level I -II
* Those children should understand and follow simple orders.

Exclusion Criteria:

* Child having any fixed deformity of both hands and feet.
* Having hearing or visual disability
* Having infectious disease or any open wound
* Seizures
* Other spinal deformities
* Any fracture
* Unstable cardiac status, Fever greater than 38 degrees Celsius, Any chest infection

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Trunk control measure scale | 6 weeks
  Trunk control measuring scale TCMS:
  Trunk control measuring scale is highly reliable in children with various neuromuscular disorders .It is reliable for children 5 years and older. TCMS consist of static and dynamic
  sitting balance, the latter is divided into selective movement control and dynamic reaching.
  TCMS is a valid and reliable tool for assessing the trunk control in children and youth with CP. The TCMS scale assesses seated trunk control in three dimensions. The maximum score is 58 points where 20 points correspond to static balance, 28 to selective movement control and 10 to the ability to perform dynamic reaching. The items are scored 0 to 3 with 0 being the inability to perform the task and 3 being the complete task performance.
Timed Up and Go test | 6 weeks
  Timed Up and Go test (TUG)
  It is a performance measure designed to assess the speed of a functional walk. It included stand up, walk 3 min, turn around, walk back, and sit down .It assesses lower limb mobility and function. The TUG test is reliable and responsive measure of balance and mobility for children with CP between 3 and 10 years of age and with GMFM level I- III

CONTACTS AND LOCATIONS:
Overall Officials: Maidah Aiman, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Germain AM, Blackmore AM, Gibson N, Newell B, Williams SA. Effects of Adaptive Bungee Trampolining for Children With Cerebral Palsy: A Single-Subject Study. Pediatr Phys Ther. 2019 Apr;31(2):165-174. doi: 10.1097/PEP.0000000000000584. PMID 30865143